CLINICAL TRIAL: NCT04415190
Title: Multicenter Retrospective Study Evaluating the Impact of Early Palliative Care on the Survival of Patients With Locally Advanced and / or Metastatic Cholangiocarcinoma (CCK)
Brief Title: the Impact of Early Palliative Care on the Survival of Locally Advanced and / or Metastatic Cholangiocarcinoma Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Anthony LOPEZ, Dr Lopez, MCU, Central Hospital, Nancy, France
Other Study IDs: 2019PI274
Record Dates: First submitted 2020-05-29; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cholangiocarcinoma with early palliative care
  Interventions: Other: early palliative care
- cholangiocarcinoma without early palliative care

INTERVENTIONS:
Other: early palliative care — early palliative care
  Groups: cholangiocarcinoma with early palliative care

SUMMARY:
The prognosis for cholangiocarcinoma is bad. Potentially, early management by a palliative care team could increase overall survival. We will also assess whether early management by a palliative care team could impact progression-free survival, the place of death and the date of the last chemotherapy, in particular to avoid unnecessary chemotherapy cures in an imminent end of life

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years old
* intra- or extra-hepatic CCK or histologically proven vesicular adenocarcinoma
* Locally advanced and / or metastatic disease from the start or recurrent
* Initial diagnosis or recurrence between 1/01/2013 and 31/12/2019

Exclusion Criteria:

* <18 years old
* death less than one week after the diagnostic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cholangiocarcinoma metastatic or locally advanced
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Global survival | baseline
  Global survival from the diagnosis (to the death or because of lost to follow up)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Lopez, Principal Investigator — CHRU Nancy
Locations (1):
- Lopez, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided